CLINICAL TRIAL: NCT01607541
Title: Peer-driven Intervention to Seek, Test & Treat Heterosexuals at High Risk for HIV
Acronym: BCAP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R11-01257; R01DA032083 (NIH)
Record Dates: First submitted 2012-05-23; First posted 2012-05-30 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2016-06

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; vulnerable populations; heterosexuals at high risk; peer-driven intervention; tailored intervention; African-American; Latino/Hispanic; Seek, test, treat, and retain (STTR)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer-driven intervention (Experimental): The PDI entails structured intervention sessions including a computerized "CARE for Prevention" tool and HIV pre-test and post-test counseling, the opportunity to educate three peers on core education messages, and navigation for those HIV infected (if HIV-negative: total 3.5 hours of facilitated/computer intervention activities, plus peer education experiences; if HIV-positive: 5 hrs facilitated/computer activities, plus peer education experiences and six months of navigation)
  Interventions: Behavioral: BCAP peer-driven intervention (PDI)
- Control (Active Comparator): The control arm will receive a time- and attention-matched HIV counseling and testing intervention and for those found HIV-infected, an appointment with HIV services and reminders, the current standard of care.
  Interventions: Behavioral: Control intervention

INTERVENTIONS:
Behavioral: BCAP peer-driven intervention (PDI) — The Brooklyn Community Action Project (BCAP) PDI entails structured sessions including the computerized "CARE for Prevention" tool, 3 peer education experiences, and 6 months of navigation for those HIV infected (if HIV-negative: total 3.5 hours of facilitated/computer intervention activities, plus peer education experiences; if HIV-positive: 5 hrs facilitated/computer activities, plus peer education experiences and navigation).
  Other Names: Brooklyn Community Action Project (BCAP) PDI
  Arms: Peer-driven intervention
Behavioral: Control intervention — The control arm will receive a time- and attention-matched HIV counseling and testing intervention and for those found HIV-infected, an appointment with HIV services and reminders, the current standard of care.
  Arms: Control

SUMMARY:
Approximately 21% of HIV infections in the U.S. are undiagnosed, but only about 40% of all adults have been tested. Thus, late diagnosis of HIV is common, and, furthermore, treatment delays and disruptions are widespread. Heterosexuals at high risk (HHR) are significantly less likely to test for HIV, are more likely to be diagnosed with HIV late, and experience serious barriers to entering care compared to other groups. The investigators research team has studied HHR in New York City (NYC) as part of the CDC's National HIV Behavioral Surveillance (NHBS) studies. The investigators found an HIV prevalence rate of 7.4% among HHR in NYC, and only 6% of these infections had been previously diagnosed. Further, in central Brooklyn, 10% were newly diagnosed with HIV. The proposed study will use NHBS methodology to target HHR in central Brooklyn.

The primary goal of the proposed study is to evaluate the efficacy of a peer-driven intervention (PDI) to seek, test, treat and retain HHR. The investigators will also compare the effectiveness of two sampling methods to reach HHR: Respondent-driven sampling (a peer-based approach) versus venue-based sampling (a location-based approach).

The two main study hypotheses are:

(H1): Participants recruited by respondent-driven sampling (RDS) will be more likely to test positive for HIV compared to those recruited via venue-based sampling (VBS).

H2): Participants in the "Test and Treat: phase of the peer-driven intervention (all of whom will be HIV-infected) will show a shorter time to an HIV clinical appointment, a shorter time to starting HIV medication (when medically indicated), higher rates of viral load suppression, and higher rates of retention in care compared to those in the control arm.

DETAILED DESCRIPTION:
Approximately 21% of HIV infections in the U.S. are undiagnosed, but only about 40% of all adults have been tested. Thus, late diagnosis of HIV is common, and, furthermore, treatment delays and disruptions are widespread. Heterosexuals at high risk (HHR) are significantly less likely to test for HIV, are more likely to be diagnosed with HIV late, and experience serious barriers to entering care compared to other groups. Our research team has studied HHR in New York City (NYC) as part of the CDC's National HIV Behavioral Surveillance (NHBS) studies. The investigators found an HIV prevalence rate of 7.4% among HHR in NYC, and only 6% of these infections had been previously diagnosed. Further, in central Brooklyn, 10% were newly diagnosed with HIV. The proposed study will use NHBS methodology to target HHR. Reduced rates of HIV testing and treatment among HHR are due to structural (e.g., poor access), social (e.g., peer norms), and individual-level (e.g., low perceived risk) barriers. Thus active recruitment approaches modeled after NHBS are needed to overcome structural barriers, and peer-delivered interventions effectively reduce individual and social barriers to testing and treatment. The primary goal of the proposed study is to evaluate the efficacy of a multi-level enhanced peer-driven intervention (PDI) to seek, test, treat and retain HHR. The enhanced PDI is tailored specifically for HHR and includes computerized, navigation, and peer-delivered components to enhance future sustainability. The design of the intervention is guided by the Theories of Triadic Influence and Normative Regulation. Similar to NHBS, the enhanced PDI will use respondent-driven sampling (RDS). NHBS protocols use both venue-based sampling (VBS) and RDS for reaching populations at high risk. However, VBS and RDS have not yet been directly compared in terms of their yield of undiagnosed HIV infections. Thus the specific aims of this five-year proposed study are to: (1) compare the yield and efficiency of RDS and VBS to identify undiagnosed HIV infection among HHR; (2) measure the efficacy of an enhanced PDI compared to a control in terms of time to HIV care and HAART initiation, viral load suppression, and retention among those newly-diagnosed; (3) examine whether the effects of the PDI on HIV health/treatment outcomes are mediated by changes in individual (e.g., perceived risk), social (e.g., peer norms), and structural influences (e.g., enhanced access), and/or whether other factors (e.g., substance use) moderate its effects; and (4) to project the costs and cost-effectiveness of RDS vs. VBS and PDI.

The investigators will conduct the enhanced PDI (N=3000) in central Brooklyn, a location hyperendemic for HIV and where HHR experience poor access to testing and treatment. Simultaneously, VBS (N=400) will be undertaken in central Brooklyn. The proposed study complements local and national HIV prevention initiatives and is designed to contribute an efficient, innovative, and sustainable multi-level recruitment approach and intervention to the HIV prevention portfolio. The vast majority of HHR are African-American or Latino; therefore the proposed study may also impact racial/ethnic disparities in HIV/AIDS.

The study's main hypotheses are as follows:

(H1): Compared with venue-based sampling (VBS), and controlling for potential differences on key sociodemographic characteristics across the samples, participants recruited by respondent-driven sampling (RDS) will be more likely to test positive for HIV for the first time.

H2): Participants in the Test and Treat Phase of the BCAP PDI's intervention arm (all of whom will be HIV-infected) will evidence a shorter time to an HIV clinical appointment, a shorter time to initiating HAART (when medically indicated), higher rates of viral load suppression, and higher rates of retention in care compared to those in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-60 years
* sexually active (vaginal, anal) with at least 1 opposite sex partner within the previous year
* reside in the central Brooklyn HRA defined in the Development Phase
* African-American or Latino/Hispanic race/ethnicity
* comprehend English or Spanish
* willing to provide locator information
* willing to try to recruit peers
* not actively psychotic based on valid screening instrument
* not a participant in the two past NHBS studies with HHR (called HET1/HET2); not enrolled already in VBS or PDI/RDS in this study
* willing to be randomly assigned to intervention arm (initial seeds only, for PDI component)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3400 (Actual)
Dates: Start 2012-04; Primary Completion 2015-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
proportion of newly diagnosed HIV infections | 2 months post-baseline
time to HIV clinical appointment | 12-months post intervention
time to initiation of HAART if medically indicated | 12-months post intervention
viral load suppression | 12-months post intervention
retention in care | 12 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marya Gwadz, PhD, Principal Investigator — New York University
Locations (1):
- New York University College of Nursing, New York, New York, United States

REFERENCES:
- [Derived] Gwadz M, Cleland CM, Hagan H, Jenness S, Kutnick A, Leonard NR, Applegate E, Ritchie AS, Banfield A, Belkin M, Cross B, Del Olmo M, Ha K, Martinez BY, McCright-Gill T, Swain QL, Perlman DC, Kurth AE; BCAP Collaborative Research Team. Strategies to uncover undiagnosed HIV infection among heterosexuals at high risk and link them to HIV care with high retention: a "seek, test, treat, and retain" study. BMC Public Health. 2015 May 10;15:481. doi: 10.1186/s12889-015-1816-0. PMID 25958200